CLINICAL TRIAL: NCT04257838
Title: Monitoring of Piperacillin-Tazobactam and Meropenem Plasmatic Levels in Critical Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-MER-2019-01
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic Shock; Piperacillin-Tazobactam; Meropenem; Plasmatic Levels; Critical Patients; Dose adjustment
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Piperacillin; Tazobactam; Meropenem

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Piperacillin-Tazobactam or Meropenem Cohort: Patients hospitalized for sepsis or septic shock that are treated with Piperacillin-Tazobactam or Meropenem and meet all the inclusion criteria and none of the exclusion criteria.
  Interventions: Drug: Piperacillin/tazobactam or Meropenem

INTERVENTIONS:
Drug: Piperacillin/tazobactam or Meropenem — The plasmatic levels determinations will always be made in state of equilibrium (after the fourth dose) and two samples will be collected:
  1. Just before the antibiotic infusion (T0)
  2. In the midpoint of time (T50). If the antibiotic is administered every 8 hours this determination will be made at 4 hours. If the antibiotic is administered every 6 hours, the determination will be made at 3 hours.
  A second complete determination will be made (before the infusion, in the midpoint of time and before the next dose) after the administration of 4 doses as long as a posology modification is made as a consequence of the information received from the plasmatic levels.

SUMMARY:
The aim of this study is to establish the Piperacillin-Tazobactam and Meropenem Plasmatic Levels to know if it´s necessary to make some adjustment in the recommended dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old.
* Hospitalized in the Intense Care Unit.
* Patients treated with Piperacillin-Tazobactam or Meropenem.
* Septic shock.
* Renal hyper clearance.
* Gram-negative bacillary bacteremia.
* Continuous renal replacement technique.
* ECMO.
* Obesity (BMI> 40).

Exclusion Criteria:

* Patients under 18 years old.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock who are being treated with Meropenem or Piperacillin-Tazobactam and meet the following criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy . | Up to 12 months after the antibiotic administration
  The chosen efficiency parameter is that 100 % of the time the concentration remains 4 times above the minimum inhibitory concentration (MIC), the exact minimum inhibitory concentration (MIC) of the used antibiotic will be determined by E-test by the Microbiology Service which means that the seric concentrations asociated with the maximum therapeutic efficacy are:
  * For Meropenem 2mg/dl, which means reaching a concentration in T0 >8 mg/dL.
  * For Piperacillin-Tazobactam 16 mg/dL, which means reaching a concentration in T0 >64 mg/dL.

SECONDARY OUTCOMES:
Evaluate if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy in patients with renal hyper clearance. | Up to 12 months after the antibiotic administration
  The seric concentrations asociated with the maximum therapeutic efficacy are the same as the described for the description of the Primary Outcome Measure and it´s considered that a patient has renal hyper clearance when they have a creatinine clearance above 130 ml/min.
Evaluate if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy in patients with Gram-negative bacillary bacteremia. | Up to 12 months after the antibiotic administration
  The seric concentrations asociated with the maximum therapeutic efficacy are the same as the described for the description of the Primary Outcome Measure and it´s considered that a patient has Gram-negative bacillary bacteremia when the bloodstream is invaded by Gram-negative bacillary which is diagnosed by blood culture.
Evaluate if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy in patients with continuous renal replacement technique. | Up to 12 months after the antibiotic administration
  The seric concentrations asociated with the maximum therapeutic efficacy are the same as the described for the description of the Primary Outcome Measure and a patient with continuous renal replacement technique, has its blood purified extracorporeally, replacing the renal function continuously 24 hours of the day.
Evaluate if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy in patients with ExtraCorporeal Membrane Oxygenation. | Up to 12 months after the antibiotic administration
  The seric concentrations asociated with the maximum therapeutic efficacy are the same as the described for the description of the Primary Outcome Measure and a patient with ExtraCorporeal Membrane Oxygenation has a short-term extracorporeal circulatory and respiratory mechanical assistance system.
Evaluate if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy in patients with morbid obesity. | Up to 12 months after the antibiotic administration
  The seric concentrations asociated with the maximum therapeutic efficacy are the same as the described for the description of the Primary Outcome Measure and it´s considered that a patient has morbid obesity when it´s BMI (body mass index) is above 40.
Determine in the total cohort if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy. | Up to 12 months after the antibiotic administration
  Determine in the total cohort if with the currently recommended dose regimen for Piperacillin-Tazobactam and Meropenem are achieved the seric concentrations asociated with the maximum therapeutic efficacy.
Determine the association between the supra-therapeutic levels and the appearance of toxicity. | Up to 12 months after the antibiotic administration
  Determination of if there´s an association between the antibiotics supra-therapeutic levels and the toxicity appearance.

CONTACTS AND LOCATIONS:
Overall Officials: José Garnacho Montero, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain